CLINICAL TRIAL: NCT03185364
Title: The Safety and Efficiency of Sildenafil in the Treatment of Severe Post-capillary Pulmonary Hypertension Caused by COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jianguo He, Chief of Pulmonary Vascular Disease Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016YFC1304401B
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: COPD; Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: 23 patients use placebo and 23 patients use sidenafil for 12 weeks' treatment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Sildenafil Citrate, 20mg, tid for 12 weeks
  Interventions: Drug: Sildenafil Citrate
- Control group (Placebo Comparator): placebo oral tablet, 12 weeks
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Sildenafil Citrate — sildenafil treatment for 12 weeks, monitoring blood pressure and other adverse events
  Arms: Interventional group
Drug: Placebo Oral Tablet — placebos treatment for 12 weeks
  Arms: Control group

SUMMARY:
Over half of chronic obstructive pulmonary disease (COPD) patients develop pulmonary hypertension. The current therapy focuses only on the basic disease and there are a lot of controversies about the use of PAH target therapy in group 3 pulmonary hypertension. Our study is to explore whether sildenafil, a pulmonary arterial hypertension (PAH) target drug, could be efficient and safe in improving symptoms and survival of severe pulmonary hypertension caused by COPD.

ELIGIBILITY:
Inclusion Criteria:

* Stable for over 1 month
* mean pulmonary artery pressure ≥35mmHg, pulmonary wedge pressure≤ 15mmHg
* never received target therapy before

Exclusion Criteria:

* Patients with other serious respiratory diseases
* Patients with pulmonary hypertension other than group 3
* Patients with right heart hypertrophy or dysfunction not caused by chronic obstructive pulmonary diseases
* Patients with limited life expectancy
* Patients with history of tracheal intubation or stoke, acute coronary syndrome in 6 months
* Psychopath or addict
* Nonstable patients with type Ⅰor Ⅱ respiratory failure
* Patients with contraindication for sildenafil
* Patients in pregnancy or breastfeeding

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
pulmonary artery pressure | 12 weeks
  pressure in mmHg
pulmonary vascular resistance | 12 weeks
  woods

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided